CLINICAL TRIAL: NCT02823938
Title: Sample Analysis Generalist Beneficiaries of Health Insurance From 2004 to 2014
Brief Title: DRUG EXPOSURE AND RISK OF DEMENTIA
Acronym: EXMEDEM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9641
Record Dates: First submitted 2016-06-30; First posted 2016-07-06 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Affiliated to the General Scheme

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: existing database on data collection. — This is an observational study on an existing database.

SUMMARY:
In France, a person consumes an average of 48 boxes of medicines per year (ANSM 2012). Among these substances, some, not prescribed in an indication related to cognitive function, however, will influence thereon.

Several drug candidates with potential preventive effects have already been explored with little success (statins, antihypertensives, NSAIDs, aspirin, steroid hormones). Other studies have suggested the existence of deleterious cognitive effects of certain substances (benzodiazepines, anticholinergics, anti-cancer chemotherapy). However, only the effects of a limited number of drugs were analyzed, and most drugs have not been specific study in epidemiology.

The study of this research theme has often been restricted by the limited size of the cohort of staff, not allowing the study of sometimes rare drug exposures, and poverty of the information collected on drug exposures. Thus, most studies focuses on families of molecules among the most prescribed. In addition, we now know that the pathophysiological process underlying Alzheimer's disease (representing 2/3 of dementia), actually begins more than 10 years before the diagnosis of dementia. It is therefore essential to have a setback of several years between drug exposure and diagnosis of dementia to assess their role in the genesis and evolution of the disease.

The Generalist Sample Beneficiaries (EGB) is a database containing data of health insurance and those of medicalization program of information systems (PMSI) for a sample of 550 000 subjects enrolled in the general scheme of the insurance since 2004 and followed for a period of 20 years.

DETAILED DESCRIPTION:
In France, a person consumes an average of 48 boxes of medicines per year (ANSM 2012). Among these substances, some, not prescribed in an indication related to cognitive function, however, will influence thereon.

Several drug candidates with potential preventive effects have already been explored with little success (statins, antihypertensives, NSAIDs, aspirin, steroid hormones). Other studies have suggested the existence of deleterious cognitive effects of certain substances (benzodiazepines, anticholinergics, anti-cancer chemotherapy). However, only the effects of a limited number of drugs were analyzed, and most drugs have not been specific study in epidemiology.

The study of this research theme has often been restricted by the limited size of the cohort of staff, not allowing the study of sometimes rare drug exposures, and poverty of the information collected on drug exposures. Thus, most studies focuses on families of molecules among the most prescribed. In addition, we now know that the pathophysiological process underlying Alzheimer's disease (representing 2/3 of dementia), actually begins more than 10 years before the diagnosis of dementia. It is therefore essential to have a setback of several years between drug exposure and diagnosis of dementia to assess their role in the genesis and evolution of the disease.

The Generalist Sample Beneficiaries (EGB) is a database containing data of health insurance and those of medicalization program of information systems (PMSI) for a sample of 550 000 subjects enrolled in the general scheme of the insurance since 2004 and followed for a period of 20 years.

ELIGIBILITY:
Inclusion Criteria:

* from over 60 and under 85 years in 2011,
* Affiliated to the general scheme and present in the base of the EGB since 2004
* Not diagnosed as demented before 2011

Exclusion Criteria:

* NA

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will include in our analyzes all subjects over 60 and under 85 years in 2011 and affiliated to the general scheme present in the base of the EGB since 2004, undiagnosed dementia as before 2011, approximately 120,000 subjects.
Sampling Method: Probability Sample
Enrollment: 120000 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
drug exposures | 1 year
  drug exposures (grouped by therapeutic class and / or analyzed molecule by molecule) in 2004-2005-2006

SECONDARY OUTCOMES:
dementia occurred | 1 year
  dementia occurred in 2011, 2012, 2013 or 2014

CONTACTS AND LOCATIONS:
Overall Officials: Thibault MURA, Study Director — UH MONTPELLIER
Locations (1):
- UHMontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC